CLINICAL TRIAL: NCT05323474
Title: Optimized Rehabilitation After Anterior Cruciate Ligament Reconstruction at the First Step of Return to Sport
Brief Title: Optimized Rehabilitation After Anterior Cruciate Ligament Before Returning to Sport
Acronym: ORACL-Run
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20PH282; 2022-A00287-36 (Other: ANSM)
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Ligament Knee Injury; Anterior Cruciate Ligament Rupture
Keywords: Physiotherapy; Rehabilitation; Orthopedic surgery; Knee joint; Ligament; Anterior Cruciate Ligament Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard rehabilitation (Experimental): Classical rehabilitation carried out by a physiotherapist with an evaluation at 6 months post-surgery to authorize the return to sport.
  Interventions: Other: Usual rehabilitation
- Optimized rehabilitation (Active Comparator): Classical rehabilitation carried out by a physiotherapist + expert physiotherapist performing monthly clinical and functional assessments with recommendations for exercises and running program sent to the physiotherapist.
  Interventions: Other: Rehabilitation optimized

INTERVENTIONS:
Other: Usual rehabilitation — Usual rehabilitation according to the practice of the "Haute Autorité de Santé" (HAS)
  Arms: Standard rehabilitation
Other: Rehabilitation optimized — Rehabilitation optimized according to the study protocol
  Arms: Optimized rehabilitation

SUMMARY:
Following reconstruction of the anterior cruciate ligament (ACL), a standardized rehabilitation protocol is carried out by a physiotherapist. In France, a well-established rehabilitation consensus guides the first phase of 3 months postoperatively and patient compliance is generally excellent. The next phase should allow a return to sport (RTS) following a continuum depending on the objectives of the sport's patient, starting with a return to running activities (RTR) and a preparatory phase for a RTS which may be authorized at 6 months post-op.

This multicentre randomized control trial aims to evaluate the effectiveness of an individualized and optimized rehabilitation program guided by monthly assessments carried out by physiotherapists from the 3rd to the 6th month postoperatively to reduce the risk of new ACL injuries (operated or healthy knee), compared to standard management.

DETAILED DESCRIPTION:
Each year more than 40,000 surgical reconstructions of the anterior cruciate ligament (ACL) by ligamentoplasty are performed in France; the rupture being most often the result of sports practice. Following this surgical reconstruction of the ACL, a standardized rehabilitation protocol is carried out by a masseur-physiotherapist. A well-established rehabilitative consensus guides the first phase of the 3 months post-operative and patient compliance is generally excellent. The next phase should allow the return to sport (RTS) by following a continuum according to the objectives of the athlete patient. In this continuum, authors distinguish the return to sports activities in the axis, such as running (RTS1), preparing the return to training (RTS2), and much later will be done by the return to competition (RTS3).RTS2, which is probably the most delicate stage due to the highly variable progression from one patient to another, is generally allowed from the 6th month post-operative, after the realization and validation of a battery of tests assessing the athlete's ability to resume training.Despite this precaution, there is a major risk of new injury (20%), especially in the contralateral knee (12%) requiring new, longer, more restrictive rehabilitation care with an additional 3 to 12 months' incapacity for work or sport.. As the risk of "re-injury" of the knee seems independent of the surgical technique used and the first 3 months of rehabilitation, the rehabilitative management of this phase of 3 to 6 months post-operative appears decisive in the prevention of a new injury. The return to running (in the RTS1) therefore seems a major objective for rehabilitation and will build the necessary foundation for the resumption of the patient's favorite sport, RTS2. However, to allow the return to running, no objective criteria have been validated to date and no consensus is identifiable in the scientific literature. It is the same for his preparation and the gradual resumption of running. Thus, an optimized rehabilitation between the 3rd and 6th month, based on objective evaluations of the patient's functional abilities allowing personalized rehabilitation, including guided and individualized running training, could reduce the risk of new ACL injuries (operated or healthy knee) by better preparing the patient for RTS2: the return to his favorite sport

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to the French Social Security system
* Patient who has had an ACL reconstruction regardless of the standard surgical technique used
* Patient with a sports activity, pivot and/or contact (e.g. soccer, basketball, handball, rugby, judo...) and practiced in competition (Tegner sports activity scores >7 and Marx scores >11 before the accident.
* Patient wishing to return to competitive sport
* Consent signed by the patient

Exclusion Criteria:

* Contralateral or bilateral involvement or operated on for a re-injury of the ACL
* Patients with a medical contraindication to the performance of one of the tests
* Patients suffering from a neurological (motor and/or sensitive), vestibular or rheumatic pathology
* Patient performing rehabilitation with a physiotherapist who does not wish to participate in the study.
* Pregnant or breastfeeding woman
* Patient under guardianship or curators

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 432 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one new ACL injury | At 24 months post surgery
  A re-rupture of the operated ACL or a rupture on the contralateral side, objectified by a Lachman test performed with the absence of a "firm" stop, and a difference in laxity measured with an arthrometer ( >3 mm for the KT-1000 ™ or >3 mm for the GNRB® or >5 mm for the Telos™ ) and by an MRI diagnosing an ACL rupture.

SECONDARY OUTCOMES:
Number of patients meeting all the criteria necessary for authorization to return to their usual sports activities | At 6 months post surgery
  The criteria are :
  * Recovery of symmetry of muscle strength of the Quadriceps with a Limb Symmetry Index (LSI) > 90%
  * International Knee Documentation Committee (IKDC) score > the 15th percentile of subjects of the same age
  * Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) score >56
Number of patients with at least one post-surgical complication | At 24 months post surgery
  Post-surgical complications are :
  * residual flexion (>5°) measured by goniometric joint assessment,
  * knee flexion deficit (>10°) measured by goniometric joint assessment,
  * Cyclops syndrome as measured by Magnetic resonance imaging (MRI),
  * secondary symptomatic meniscal lesions objectified by a clinical examination performed by a physician and an MRI,
  * Myo-aponeurotic lesions objectified by a clinical examination performed by a physician and medical imaging (MRI or ultrasound).
Number of patients with <10% asymmetry in running biomechanical parameters | At 6 month post surgery
  Asymmetry <10% in biomechanical running parameters (stride length or stiffness coefficient of each lower limb)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas NERI, MD, Study Chair — CHU DE SAINT-ETIENNE; Grégory MOREL, Physio, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (7):
- France (6):
  - Medipole de Savoie, Challes-les-Eaux
  - Clinique de Domont Ortholab, Domont
  - Centre Hospitalier de Firminy, Firminy
  - Clinique de La Sauvegarde, Lyon
  - Hopital de La Croix Rousse, Lyon
  - CHU de Saint-Etienne, Saint-Etienne
- Hôpital de la Tour, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No